CLINICAL TRIAL: NCT00291720
Title: Is Spironolactone Safe and Effective in the Treatment of Cardiovascular Disease in Mild Chronic Renal Failure?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Birmingham (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Research & Development Office, University Hospital Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPK2749; 04/Q2707/294
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Chronic Kidney Disease; Cardiovascular Disease
Keywords: Aldosterone; Spironolactone; Chronic Kidney Disease; Arterial Stiffness
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spironolactone (Active Comparator): 25mg spironolactone daily
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): matching placebo medication for the control group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — All patients receive a 4 week open labeled run in phase of 25mg spironolactone daily after which they are randomized to continue or receive matched placebo for 8 months.
  Arms: Spironolactone
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
Patients with kidney failure have a poor survival rate that is due to a much higher than average rate of heart and vascular disease. The reason that kidney failure causes heart disease is unknown but recent research suggests that a hormone called aldosterone, which is increased in patients with kidney disease may damage the heart and blood vessels.

The investigators propose, using a randomized blinded trial, to find out whether drugs that inhibit the actions of aldosterone have beneficial effects on the cardiovascular system in patients with kidney failure

DETAILED DESCRIPTION:
Cardiovascular disease leads to the death of over half of patients with chronic renal failure (CRF) but the causes of this 'vasculopathy' remain unknown. Aldosterone is present in the circulation of renal failure patients at high levels and is known to exert damaging effects upon the myocardium, vasculature and autonomic nervous system. Patients will be randomised to determine the effect of chronic treatment with an aldosterone receptor inhibitor on left ventricular mass, diastolic function, arterial stiffness and autonomic function. All of these endpoints are predictors of mortality so that the results of this study may yield information of prognostic value and provide the basis for a future mortality study.

Premature cardiovascular disease is the leading cause of mortality in CRF accounting for approximately 60% of deaths. Across the age range, cardiovascular mortality is 10 and 20 times greater than controls but in young patients the relative risk is extreme. Dialysis patients under the age of 45 have over 100 times the risk of cardiovascular death than the control population. An increased risk is also present in patients with mild renal impairment, which has been estimated to occur in approximately 8% of the population. Thus, renal dysfunction is a potentially important risk factor for coronary artery disease in the general population. This study builds upon previous and current BHF funded work by Dr Townend and colleagues in Birmingham (PG97/162 and PG02/153) which has resulted in a number of publications in the area of cardiovascular disease in renal failure but takes a new approach examining the potential role of aldosterone in renal 'vasculopathy'.

Pathophysiology of myocardial and vascular disease in chronic renal failure:

The main pathological features of the cardiovascular system of patients with renal failure are:

1. LVH often accompanied by systolic and diastolic dysfunction.
2. Arterial wall thickening, stiffening and calcification (arteriosclerosis).
3. Coronary and peripheral artery atherosclerosis.

The pathophysiology of cardiovascular disease in renal failure is poorly understood but as renal function declines, a range of abnormalities occur that may exert adverse effects upon the cardiovascular system. Hypertension, chronic anaemia and activation of the renin-angiotensin-aldosterone system (RAAS) and sympathetic nervous system all contribute to the development of myocardial hypertrophy and fibrosis. The same abnormalities may also lead to muscular hypertrophy and fibrosis of the arterial walls including the aorta. In combination with an increase in extracellular matrix, loss of elastic fibres and diffuse medial calcification, the arterial wall changes lead to arterial 'stiffening'. In addition to these adverse haemodynamic and structural changes, endothelial injury, the first physiological manifestation of atherosclerosis, occurs early in the course of renal failure.

Hypertension, anaemia, chronic inflammation, an atherogenic lipid profile, diabetes and less certainly hyperhomocysteinaemia and abnormal calcium/phosphate metabolism are possible causes of endothelial injury and recent evidence suggests that to this list should now be added angiotensin II (ANG II) and aldosterone.

Aldosterone and cardiovascular disease: The fundamental role of the RAAS in cardiovascular disease is apparent from the results of many large ACE inhibitor trials. In patients with chronic heart failure and in those with or at high risk of coronary artery disease, ACE inhibitors improve survival, functional status and hospitalisation. These beneficial effects have been attributed to prevention of the multiple adverse effects of ANG II. More recently, evidence has accumulated in support of an important role for aldosterone.

The persistent elevation of ANG II and aldosterone concentrations during ACE inhibitor therapy is often termed 'escape'. Aldosterone secretion from the adrenal cortex persists in response to ANG II (produced by the non ACE enzymatic conversions of ANG I) and a rise in plasma potassium. Comparison of the effects of adding ANG II receptor blockers (ARB) and aldosterone receptor antagonists to ACE inhibitors in heart failure trials suggests that it is aldosterone escape that exerts the greater pathophysiological effects. In ValHeFT the addition of valsartan to ACE inhibitor therapy had no detectable effect on mortality. In both the RALES and EPHESUS trials however, mortality was significantly reduced by the addition of spironolactone (RALES) or eplerenone (EPHESUS) to standard therapy including ACE inhibitors.

Aldosterone is synthesised in numerous tissues and mineralocorticoid receptors are present in the brain, heart and blood vessels as well as the kidney. In addition to its physiological role in the kidney aldosterone exerts several pathological actions on the cardiovascular system:

1. Endothelial dysfunction: The administration of aldosterone and sodium to rats results in transmural coronary arterial inflammation with monocyte and macrophage infiltration and the expression of inflammatory markers such as COX-2, MCP-1 and VCAM-1. The administration of an aldosterone antagonist markedly reduced this inflammatory response. Although a similar response occurred with infusion of ANG II, this was in part dependent on aldosterone synthesis as it was reduced by adrenalectomy but restored by aldosterone infusion. In vitro, vascular endothelial fibrinolysis is inhibited by aldosterone as a result of an increase in plasminogen activator inhibitor (PAI-1). In humans, primary hyperaldosteronism is associated with endothelial dysfunction compared to normal and hypertensive controls. In patients with chronic heart failure, aldosterone receptor blockade with spironolactone results in significant improvement in endothelial dependent vasodilatation and vascular nitric oxide bioactivity.
2. Myocardial and vascular hypertrophy and fibrosis: Aldosterone appears to cause myocardial and vascular injury independently of effects on blood pressure. Chronic aldosterone infusion and sodium loading resulted in myocardial fibrosis and ventricular hypertrophy in rats. Treatment with aldosterone receptor antagonists prevented aortic and myocardial fibrosis in rat models of hypertension even in the absence of blood pressure lowering. In addition, in aldosterone treated stroke-prone hypertensive rats, spironolactone exerted a powerful protective effect against the development of nephrosclerotic and cerebrovascular lesions. The mechanisms of action of aldosterone may include upregulation of AT1 receptors, direct effects on fibroblast collagen synthesis and possibly decreased matrix metallo-proteinase secretion. In humans, aldosterone concentrations have been correlated with mortality in chronic heart failure, with the severity of LVH in non-diabetic renal failure and hypertension and negatively with carotid artery compliance in hypertension. When added to ACE inhibitors, treatment with aldosterone receptor antagonists further reduces LVH in both hypertension and heart failure. Myocardial collagen turnover (a marker for fibrosis) was significantly reduced by spironolactone in the RALES study and the fall in the marker of this index was related to the mortality benefit.
3. Autonomic dysfunction: Like heart failure, renal failure is characterised by autonomic dysfunction manifest by high resting sympathetic tone, impaired vagal control and reduced baroreflex sensitivity. The prognostic significance of autonomic dysfunction is not established for renal failure, but in chronic heart failure, the degree of dysfunction, measured by techniques such as heart rate variability, is a powerful and independent marker of prognosis. This evidence, coupled with the efficacy of beta-blocker therapy in heart failure, suggests that autonomic dysfunction can actively contribute to mortality and cardiovascular disease progression. Aldosterone appears to increase sympathetic and reduce cardiac vagal influence. The action of the sympathetic nervous system is increased as a result of reduced uptake of noradrenaline in the myocardium. A reduction in baroreflex sensitivity in response to aldosterone infusion has been demonstrated in both animals and man and in heart failure patients, an increase in heart rate variability occurred in response to aldosterone inhibition. We have recently shown that acute aldosterone receptor inhibition results in improved HRV markers of cardiac parasympathetic control in healthy subjects.
4. Is the effect of aldosterone receptor blockade with spironolactone mediated by lowering arterial pressure? Spironolactone is now recognised as an effective anti-hypertensive agent for patients with hypertension, even when this is resistant to other drugs. It is therefore necessary to consider whether any improvements that do occur in measures such as arterial stiffness and LV mass after spironolactone might simply be due to this effect. Several lines of evidence suggest that the effects of aldosterone inhibition are independent of blood pressure. The work of Rocha et al. in experimental animals clearly showed that inhibition of myocardial and aortic fibrosis, nephrosclerotic and cerebrovascular lesions by aldosterone inhibition occurred in the absence of changes in blood pressure. In humans, in the RALES and EPHESUS studies, the mortality effects occurred in the absence of any fall in blood pressure. In patients with controlled hypertension and diabetic nephropathy, a group relevant to the work proposed in this application, high dose spironolactone treatment (100 mg per day) did not result in a fall in either systolic or diastolic blood pressure but did reduce albuminuria independently of blood pressure. Finally, Professor Struthers, a national authority on aldosterone and the cardiovascular system, has shown that in trials of spironolactone in severe heart failure and diabetes, no fall in blood pressure occurred with spironolactone suggesting that the beneficial action of spironolactone on endothelial function was not mediated by such an effect. (personal communication). Nevertheless, an effect mediated by a reduction in blood pressure cannot be excluded. In order to examine this hypothesis, we will examine the relationship between the magnitude of changes in end points and changes in blood pressure.

The renin-angiotensin-aldosterone system in chronic renal failure: The importance of the RAAS in CRF is illustrated by the efficacy of ACE inhibitors in retarding the progression of diabetic and non-diabetic renal disease. The significance of ANG II mediated renal damage was shown by the finding that combined treatment with ACE inhibitors and ARBs further slows the progression of non-diabetic renal disease compared with either agent alone.

Plasma aldosterone concentrations are increased in animal models of CRF as well as in patients with even mild renal impairment and several lines of evidence point to a major role of aldosterone in promoting progressive renal dysfunction. Observational studies in patients with primary hyperaldosteronism found the prevalence and degree of proteinuria to be greater than in patients with essential hypertension. Several experimental animal models are consistent with the concept that aldosterone can mediate renal injury. In patients with diabetic nephropathy and aldosterone escape despite ACE inhibitor therapy, aldosterone blockade significantly reduced proteinuria with no change in blood pressure. Little attention has been paid however, to the potentially beneficial effects of aldosterone antagonism on the cardiovascular system in renal failure. In a single, small uncontrolled study of 13 patients with diabetic nephropathy on established ACE inhibitor therapy, left ventricular mass index was significantly reduced after 24 weeks of treatment with spironolactone.

Left ventricular hypertrophy and arterial stiffness as endpoints in studies in chronic renal failure:

LVH: Up to 80% of patients have LVH at the start of dialysis. As with other patient groups, LVH is a powerful independent predictor of mortality in CRF and regression of LVH is associated with improved cardiac outcome.

Arterial stiffness: Large conduit arteries buffer the changes in pressure resulting from intermittent ventricular ejection. Stiffening of the arteries (loss of arterial compliance) leads to increased systolic and pulse pressure; indeed arterial stiffness is the principal determinant of pulse pressure in patients with CRF. It is also closely associated with LVH and its progression over time. Recent prospective studies have demonstrated that measures of aortic stiffness, such as aortic pulse wave velocity (PWV), and augmentation of central aortic pressure by early wave reflections (AIx), are independent and powerful predictors of all-cause and cardiovascular mortality in patients on dialysis. Indeed, in a recent prospective study, lowering aortic PWV, mainly by use of an ACE-inhibitor, was associated with an improved survival in dialysis patients. This reduction in aortic PWV was associated with a parallel reduction in mean arterial and pulse pressure in survivors. In contrast, in those who died from cardiovascular events, although mean arterial pressure was lowered to the same extent as in survivors; neither pulse pressure nor aortic PWV was significantly modified by ACE inhibition. These findings suggest that arterial stiffness is not merely a marker of arterial damage but a potentially reversible factor contributing to mortality.

In summary: Activation of the RAAS occurs early in the course of renal disease and both angiotensin and aldosterone are likely to be important factors in the pathogenesis of arterial stiffness, LVH and autonomic dysfunction. ACE inhibitors reduce arterial stiffness and LVH as well as the progression of renal dysfunction but levels of circulating aldosterone may remain high and the effects of aldosterone inhibition are unknown.

ELIGIBILITY:
Inclusion Criteria:

* Mild-moderate chronic kidney disease (glomerular filtration rate [GFR] 40-80 mls/min calculated by Cockroft-Gault equation)
* Controlled blood pressure (< 130/80 mmHg)
* On established (> 6 weeks) treatment with angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARBs).

Exclusion Criteria:

* Diabetes mellitus
* Clinical evidence of fluid overload or hypovolaemia
* Recent (< 2 months) acute myocardial infarction
* Left ventricular (LV) dysfunction (ejection fraction < 40% by echocardiography).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Changes in left ventricular mass on cardiac MRI and arterial stiffness (assessed by pulse wave velocity). | 9 months

SECONDARY OUTCOMES:
Changes in aortic distensibility and large vessel augmentation | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: John N Townend, BSc, MB ChB, MD, FRCP, FESC, Principal Investigator — University Hospital Birmingham
Locations (1):
- University Hospital Birmingham, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Background] Foley RN, Parfrey PS, Sarnak MJ. Clinical epidemiology of cardiovascular disease in chronic renal disease. Am J Kidney Dis. 1998 Nov;32(5 Suppl 3):S112-9. doi: 10.1053/ajkd.1998.v32.pm9820470. No abstract available.
- [Background] Culleton BF, Larson MG, Wilson PW, Evans JC, Parfrey PS, Levy D. Cardiovascular disease and mortality in a community-based cohort with mild renal insufficiency. Kidney Int. 1999 Dec;56(6):2214-9. doi: 10.1046/j.1523-1755.1999.00773.x. PMID 10594797
- [Background] Coulden RA, Moss H, Graves MJ, Lomas DJ, Appleton DS, Weissberg PL. High resolution magnetic resonance imaging of atherosclerosis and the response to balloon angioplasty. Heart. 2000 Feb;83(2):188-91. doi: 10.1136/heart.83.2.188. PMID 10648495
- [Background] Thambyrajah J, Landray MJ, McGlynn FJ, Jones HJ, Wheeler DC, Townend JN. Does folic acid decrease plasma homocysteine and improve endothelial function in patients with predialysis renal failure? Circulation. 2000 Aug 22;102(8):871-5. doi: 10.1161/01.cir.102.8.871. PMID 10952955
- [Background] Landray MJ, Thambyrajah J, McGlynn FJ, Jones HJ, Baigent C, Kendall MJ, Townend JN, Wheeler DC. Epidemiological evaluation of known and suspected cardiovascular risk factors in chronic renal impairment. Am J Kidney Dis. 2001 Sep;38(3):537-46. doi: 10.1053/ajkd.2001.26850. PMID 11532686
- [Background] Jardine AG, McLaughlin K. Cardiovascular complications of renal disease. Heart. 2001 Oct;86(4):459-66. doi: 10.1136/heart.86.4.459. No abstract available. PMID 11559693
- [Background] Heart Outcomes Prevention Evaluation Study Investigators; Yusuf S, Sleight P, Pogue J, Bosch J, Davies R, Dagenais G. Effects of an angiotensin-converting-enzyme inhibitor, ramipril, on cardiovascular events in high-risk patients. N Engl J Med. 2000 Jan 20;342(3):145-53. doi: 10.1056/NEJM200001203420301. PMID 10639539
- [Background] Pitt B, Zannad F, Remme WJ, Cody R, Castaigne A, Perez A, Palensky J, Wittes J. The effect of spironolactone on morbidity and mortality in patients with severe heart failure. Randomized Aldactone Evaluation Study Investigators. N Engl J Med. 1999 Sep 2;341(10):709-17. doi: 10.1056/NEJM199909023411001. PMID 10471456
- [Background] Brown NJ. Eplerenone: cardiovascular protection. Circulation. 2003 May 20;107(19):2512-8. doi: 10.1161/01.CIR.0000071081.35693.9A. PMID 12756192
- [Background] Pitt B, Remme W, Zannad F, Neaton J, Martinez F, Roniker B, Bittman R, Hurley S, Kleiman J, Gatlin M; Eplerenone Post-Acute Myocardial Infarction Heart Failure Efficacy and Survival Study Investigators. Eplerenone, a selective aldosterone blocker, in patients with left ventricular dysfunction after myocardial infarction. N Engl J Med. 2003 Apr 3;348(14):1309-21. doi: 10.1056/NEJMoa030207. Epub 2003 Mar 31. PMID 12668699
- [Background] Rocha R, Stier CT Jr, Kifor I, Ochoa-Maya MR, Rennke HG, Williams GH, Adler GK. Aldosterone: a mediator of myocardial necrosis and renal arteriopathy. Endocrinology. 2000 Oct;141(10):3871-8. doi: 10.1210/endo.141.10.7711. PMID 11014244
- [Background] Sato T, Nishinaga M, Kawamoto A, Ozawa T, Takatsuji H. Accuracy of a continuous blood pressure monitor based on arterial tonometry. Hypertension. 1993 Jun;21(6 Pt 1):866-74. doi: 10.1161/01.hyp.21.6.866. PMID 8500866
- [Background] Epstein M. Aldosterone as a determinant of cardiovascular and renal dysfunction. J R Soc Med. 2001 Aug;94(8):378-83. doi: 10.1177/014107680109400803. No abstract available. PMID 11461980
- [Background] Foley RN, Parfrey PS, Kent GM, Harnett JD, Murray DC, Barre PE. Serial change in echocardiographic parameters and cardiac failure in end-stage renal disease. J Am Soc Nephrol. 2000 May;11(5):912-916. doi: 10.1681/ASN.V115912. PMID 10770969
- [Background] London GM, Guerin AP, Marchais SJ, Pannier B, Safar ME, Day M, Metivier F. Cardiac and arterial interactions in end-stage renal disease. Kidney Int. 1996 Aug;50(2):600-8. doi: 10.1038/ki.1996.355. PMID 8840292
- [Background] Guerin AP, Blacher J, Pannier B, Marchais SJ, Safar ME, London GM. Impact of aortic stiffness attenuation on survival of patients in end-stage renal failure. Circulation. 2001 Feb 20;103(7):987-92. doi: 10.1161/01.cir.103.7.987. PMID 11181474
- [Background] Wilkinson IB, Fuchs SA, Jansen IM, Spratt JC, Murray GD, Cockcroft JR, Webb DJ. Reproducibility of pulse wave velocity and augmentation index measured by pulse wave analysis. J Hypertens. 1998 Dec;16(12 Pt 2):2079-84. doi: 10.1097/00004872-199816121-00033. PMID 9886900
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592
- [Derived] Hammer F, Edwards NC, Hughes BA, Steeds RP, Ferro CJ, Townend JN, Stewart PM. The effect of spironolactone upon corticosteroid hormone metabolism in patients with early stage chronic kidney disease. Clin Endocrinol (Oxf). 2010 Nov;73(5):566-72. doi: 10.1111/j.1365-2265.2010.03832.x. PMID 20550533
- [Derived] Edwards NC, Steeds RP, Stewart PM, Ferro CJ, Townend JN. Effect of spironolactone on left ventricular mass and aortic stiffness in early-stage chronic kidney disease: a randomized controlled trial. J Am Coll Cardiol. 2009 Aug 4;54(6):505-12. doi: 10.1016/j.jacc.2009.03.066. PMID 19643310
- [Derived] Edwards NC, Ferro CJ, Townend JN, Steeds RP. Aortic distensibility and arterial-ventricular coupling in early chronic kidney disease: a pattern resembling heart failure with preserved ejection fraction. Heart. 2008 Aug;94(8):1038-43. doi: 10.1136/hrt.2007.137539. Epub 2008 Feb 28. PMID 18308865